CLINICAL TRIAL: NCT02548078
Title: Safety and Immunogenicity Study of GSK Biologicals' Investigational Recombinant Chimpanzee Adenovirus Type 3-vectored Ebola Zaire Vaccine (GSK3390107A) in Children in Africa
Brief Title: A Study to Evaluate the Safety and Immunogenicity of a Candidate Ebola Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 202090; 2014-004714-28 (EudraCT Number)
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Results first posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-03

CONDITIONS: Virus Diseases
Keywords: Protection against Ebola Zaire virus
MeSH Terms: conditions — Virus Diseases | interventions — halofantrine; Solvents; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- GSK3390107A+Nimenrix Group (Experimental): Subjects in the GSK3390107A+Nimenrix Group received the investigational GSK3390107A vaccine at the Day 0 visit and Nimenrix at the Month 6 visit, intramuscularly into the deltoid region, or thigh region for smaller children.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' investigational recombinant chimpanzee adenovirus Type 3-vectored Ebola Zaire vaccine (ChAd3-EBO-Z) (GSK3390107A); Biological: Nimenrix powder and solvent for solution for injection in pre-filled syringe; Meningococcal group A, C, W-135 and Y conjugate vaccine
- Nimenrix+GSK3390107A Group (Experimental): Subjects in the Nimenrix +GSK3390107A Group received Nimenrix at the Day 0 visit and the investigational GSK3390107A vaccine at the Month 6 visit, intramuscularly into the deltoid region, or thigh region for smaller children.
  Interventions: Biological: GlaxoSmithKline (GSK) Biologicals' investigational recombinant chimpanzee adenovirus Type 3-vectored Ebola Zaire vaccine (ChAd3-EBO-Z) (GSK3390107A); Biological: Nimenrix powder and solvent for solution for injection in pre-filled syringe; Meningococcal group A, C, W-135 and Y conjugate vaccine

INTERVENTIONS:
Biological: GlaxoSmithKline (GSK) Biologicals' investigational recombinant chimpanzee adenovirus Type 3-vectored Ebola Zaire vaccine (ChAd3-EBO-Z) (GSK3390107A) — A single dose administered intramuscular
Biological: Nimenrix powder and solvent for solution for injection in pre-filled syringe; Meningococcal group A, C, W-135 and Y conjugate vaccine — A single dose administered intramuscular

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of a single IM dose of the GSK3390107A (ChAd3 EBO-Z) vaccine, overall and in children aged 1 to 5, 6 to 12, and 13 to 17 years, separately.

Considering the risk of exposure to Ebola and the potential (based on animal data) for the investigational GSK3390107A (ChAd3-EBO-Z) vaccine to afford at least partial protection, all children in the study will receive the investigational GSK3390107A (ChAd3 EBO-Z) vaccine. The children in the Group GSK3390107A+Nimenrix will receive the investigational GSK3390107A (ChAd3-EBO-Z) vaccine at Day 0 of the study, whereas the children in the Group Nimenrix+GSK3390107A will receive Nimenrix at Day 0 (as a control). At Month 6, the children in the Group Nimenrix+GSK3390107A will receive the investigational GSK3390107A (ChAd3-EBO-Z) vaccine (provided that no safety concerns are raised), whereas the children in the Group GSK3390107A+Nimenrix will receive Nimenrix.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s)/ legally acceptable representative(s) (LAR[s]) who, in the opinion of the Investigator, can and will comply with the requirements of the protocol (e.g. availability for Diary Card completion, return for follow-up visits, availability for clinical follow-up throughout the study period).
* Written/ thumb printed informed consent obtained from the subject' parent(s)/ LAR[s] prior to performing any study specific procedure. In addition, written/ thumb printed in-formed assent should be obtained if appropriate (from all subjects aged 13 to 17 years and from younger subjects as per local requirements).
* A male or female child aged 1 to 17 years inclusive at the time of Screening.
* Subjects with a negative RDT test for Malaria within 30 days prior to randomisation into the study.

OR Subjects with a positive RDT test for Malaria who completed antimalarial treatment at least 5 days prior to randomisation into the study.

* Healthy subjects as per Investigator judgement, as estab-lished by medical history, clinical examination and haema-tology/ biochemistry laboratory parameters screening be-fore entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche or ovariectomy.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to the Day 0 visit, and
  * has a negative pregnancy test at the Day 0 visit, and
  * has agreed to continue adequate contraception until 30 days after the Month 6 visit

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine during the period starting 30 days before the Day 0 visit, or planned use during the study period.
* Previous vaccination with an investigational EBOV or Marburg vaccine, or previous vaccination with a chim-panzee adenoviral vectored investigational vaccine.
* Known prior EBOV or SUDV disease.
* Travel to country affected by the EBOV epidemic or direct contact with person with EVD within 21 days prior to the Day 0 visit.
* History of any reaction or hypersensitivity (such as ana-phylaxis, urticaria (hives), respiratory difficulty, angioe-dema, or abdominal pain) likely to be exacerbated by any component of the study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after each vaccination visit.
* Acute or chronic illness determined by medical history, clinical examination and laboratory screening tests in-cluding, but not limited to:
* Clinically significant immunosuppressive or immunodeficient condition (e.g. clinical acquired immune deficiency syndrome [AIDS]).
* Major congenital defects.
* Malnutrition (defined as weight for age Z-score less than -3, or other clinical signs of malnutrition).
* Any clinically significant haematological or biochemical laboratory abnormality.
* Pregnant female.
* Any condition that in the Investigator's opinion may po-tentially compromise subject safety or interfere with sub-ject assessment or compliance.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Bamako, Mali
- GSK Investigational Site, Dakar, Senegal

REFERENCES:
- [Derived] Tapia MD, Sow SO, Mbaye KD, Thiongane A, Ndiaye BP, Ndour CT, Mboup S, Keshinro B, Kinge TN, Vernet G, Bigna JJ, Oguche S, Koram KA, Asante KP, Gobert P, Hogrefe WR, De Ryck I, Debois M, Bourguignon P, Jongert E, Ballou WR, Koutsoukos M, Roman F; Zaire EBola Research Alliance group. Safety, reactogenicity, and immunogenicity of a chimpanzee adenovirus vectored Ebola vaccine in children in Africa: a randomised, observer-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2020 Jun;20(6):719-730. doi: 10.1016/S1473-3099(20)30019-0. Epub 2020 Mar 19. PMID 32199492

RESULTS

PARTICIPANT FLOW:
Groups:
- Nimenrix+GSK3390107A Group: Subjects in the Nimenrix+GSK3390107A Group received Nimenrix at the Day 0 visit and the investigational GSK3390107A vaccine at the Month 6 visit, intramuscularly into the deltoid region, or thigh region for smaller children.
Period: Overall Study
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Started | 300 | 300
Completed | 295 | 294
Not Completed | 5 | 6
Not completed — Serious adverse event/Adverse event | 1 | 0
Not completed — Moved from study area | 3 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.0 (4.95) | 8.8 (5.03) | 8.90 (4.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 150 | 299
  Male | 151 | 150 | 301
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AFRICAN HERITAGE/AFRICAN AMERICAN | 300 | 300 | 600

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms, Overall
Description: Assessed solicited local symptoms included: pain and swelling at the injections site. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = crying at limb movement/spontaneous pain.Grade 3 swelling = swelling extending on a surface higher than (>) 30 millimeters (mm). Solicited local symptoms, for this endpoint, were assessed in all subjects, in both groups.
Time Frame: During a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 300 | 300
Participants
  Any Pain | 127 | 60
  Grade 3 Pain | 4 | 0
  Any Swelling | 5 | 1
  Grade 3 Swelling | 1 | 0

2. Primary Outcome: Number of Subjects With Solicited Local Symptoms, by Age Stratum
Description: Assessed solicited local symptoms included: pain and swelling at the injections site. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = crying at limb movement/spontaneous pain.Grade 3 swelling = swelling extending on a surface higher than (>) 30 millimeters (mm), for children between 1-5 years old; > 50 mm for children between 6-12 years old and >100 mm for children between 13-17 years old.
Time Frame: During a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- GSK3390107A+Nimenrix 13-17YOA Group: Sub-group of subjects from the GSK3390107A+Nimenrix Group, between and including 13 to 17 years of age (YOA), who received the investigational GSK3390107A vaccine at the Day 0 visit and Nimenrix at the Month 6 visit, intramuscularly into the deltoid region.
- Nimenrix+GSK3390107A 13-17YOA Group: Sub-group of subjects from the Nimenrix+GSK3390107A Group, between and including 13 to 17 years of age (YOA), who received Nimenrix at the Day 0 visit and the investigational GSK3390107A vaccine at the Month 6 visit, intramuscularly into the deltoid region.
- GSK3390107A+Nimenrix 6-12YOA Group: Sub-group of subjects from the GSK3390107A+Nimenrix Group, between and including 6 to 12 years of age (YOA), who received the investigational GSK3390107A vaccine at the Day 0 visit and Nimenrix at the Month 6 visit, intramuscularly into the thigh region.
- Nimenrix+GSK3390107A 6-12YOA Group: Sub-group of subjects from the Nimenrix+GSK3390107A Group, between and including 6 to 12 years of age (YOA), who received Nimenrix at the Day 0 visit and the investigational GSK3390107A vaccine at the Month 6 visit, intramuscularly into the thigh region.
- GSK3390107A+Nimenrix 1-5YOA Group: Sub-group of subjects from the GSK3390107A+Nimenrix Group, between and including 1 to 5 years of age (YOA), who received the investigational GSK3390107A vaccine at the Day 0 visit and Nimenrix at the Month 6 visit, intramuscularly into the thigh region.
- Nimenrix+GSK3390107A 1-5YOA Group: Sub-group of subjects from the Nimenrix+GSK3390107A Group, between and including 1 to 5 years of age (YOA), who received Nimenrix at the Day 0 visit and the investigational GSK3390107A vaccine at the Month 6 visit, intramuscularly into the thigh region.
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 99 | 101 | 101 | 99
Participants
  Any Pain | 31 | 14 | 41 | 23 | 55 | 23
  Grade 3 Pain | 0 | 0 | 1 | 0 | 3 | 0
  Any Swelling | 1 | 0 | 3 | 1 | 1 | 0
  Grade 3 Swelling | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Solicited General Symptoms, Overall
Description: Solicited general symptoms assessed included: fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain], headache, drowsiness, irritability/fussiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 fatigue/headache/drowsiness/gastrointestinal symptoms = fatigue/headache/drowsiness/gastrointestinal symptoms that prevented normal activity. Grade 3 fever = temperature > 39.5°C. Grade 3 irritability/fussiness = crying that couldn't be comforted. Grade 3 loss of appetite = not eating at all. Related = symptom assessed by the investigator as related to the vaccination. Solicited general symptoms, for this endpoint, were assessed in all subjects, in both groups.
Time Frame: During a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 300 | 300
Participants
  Any Fatigue | 33 | 6
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 32 | 5
  Any Fever | 95 | 28
  Grade 3 Fever | 1 | 0
  Related Fever | 89 | 26
  Any Gastrointestinal symptoms | 16 | 6
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 13 | 3
  Any Headache | 62 | 17
  Grade 3 Headache | 0 | 0
  Related Headache | 60 | 14
  Any Drowsiness | 26 | 2
  Grade 3 Drowsiness | 3 | 0
  Related Drowsiness | 26 | 1
  Any Irritability/fussiness | 10 | 2
  Grade 3 Irritability/fussiness | 4 | 0
  Related Irritability/fussiness | 10 | 2
  Any Loss of appetite | 24 | 4
  Grade 3 Loss of appetite | 3 | 0
  Related Loss of appetite | 24 | 4

4. Primary Outcome: Number of Subjects With Solicited General Symptoms, by Age Stratum
Description: Solicited general symptoms assessed included: fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain], headache, drowsiness, irritability/fussiness and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 fatigue/headache/drowsiness/gastrointestinal symptoms = fatigue/headache/drowsiness/gastrointestinal symptoms that prevented normal activity. Grade 3 fever = temperature > 39.5°C. Grade 3 irritability/fussiness = crying that couldn't be comforted. Grade 3 loss of appetite = not eating at all. Related = symptom assessed by the investigator as related to the vaccination. Solicited general symptoms, for this endpoint, were assessed in subjects aged 1-5 years, 6-12 years and 13-17 years. Symptoms with no values were not assessed for those specific age groups.
Time Frame: During a 7-day follow-up period after each vaccination (i.e. the day of vaccination and 6 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 99 | 101 | 101 | 99
Participants
  Any Fatigue: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Any Fatigue | 20 | 5 | 13 | 1 |  |
  Grade 3 Fatigue: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Grade 3 Fatigue | 0 | 0 | 0 | 0 |  |
  Related Fatigue: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Related Fatigue | 20 | 4 | 12 | 1 |  |
  Any Fever | 20 | 4 | 25 | 1 | 50 | 23
  Grade 3 Fever | 0 | 0 | 0 | 0 | 1 | 0
  Related Fever | 17 | 4 | 23 | 1 | 49 | 21
  Any Gastrointestinal symptoms: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Any Gastrointestinal symptoms | 9 | 2 | 7 | 4 |  |
  Grade 3 Gastrointestinal symptoms: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Grade 3 Gastrointestinal symptoms | 0 | 0 | 0 | 0 |  |
  Related Gastrointestinal symptoms: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Related Gastrointestinal symptoms | 8 | 0 | 5 | 3 |  |
  Any Headache: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Any Headache | 36 | 11 | 26 | 6 |  |
  Grade 3 Headache: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Grade 3 Headache | 0 | 0 | 0 | 0 |  |
  Related Headache: number analyzed (Participants) | 100 | 100 | 99 | 101 | 0 | 0
  Related Headache | 35 | 8 | 25 | 6 |  |
  Any Drowsiness: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Any Drowsiness |  |  |  |  | 26 | 2
  Grade 3 Drowsiness: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Grade 3 Drowsiness |  |  |  |  | 3 | 0
  Related Drowsiness: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Related Drowsiness |  |  |  |  | 26 | 1
  Any Irritability/fusiness: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Any Irritability/fusiness |  |  |  |  | 10 | 2
  Grade 3 Irritability/fusiness: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Grade 3 Irritability/fusiness |  |  |  |  | 4 | 0
  Related Irritability/fusiness: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Related Irritability/fusiness |  |  |  |  | 10 | 2
  Any Loss of appetite: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Any Loss of appetite |  |  |  |  | 24 | 4
  Grade 3 Loss of appetite: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Grade 3 Loss of appetite |  |  |  |  | 3 | 0
  Related Loss of appetite: number analyzed (Participants) | 0 | 0 | 0 | 0 | 101 | 99
  Related Loss of appetite |  |  |  |  | 24 | 4

5. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs), Overall
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Unsolicited adverse events, for this endpoint, were assessed in all subjects, in both groups.
Time Frame: During the 30-day follow-up period after each vaccination (i.e. the day of vaccination and 29 subsequent days)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 300 | 300
Participants | 41 | 24

6. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs), by Age Stratum
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Unsolicited AEs, for this endpoint, were assessed in subjects between 1-5 years of age, 6-12 years of age and 13-17 years of age.
Time Frame: During the 30-day follow-up period after each vaccination (i.e. the day of vaccination and 29 subsequent days)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 99 | 101 | 101 | 99
Participants | 12 | 8 | 6 | 10 | 23 | 6

7. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: Haematological parameters assessed included: complete blood count (red blood cells [RBC], neutrophils, lymphocytes, white blood cells [WBC], haemoglobin, as well as differential count and platelet count for all subjects, in both groups. Reference range indicators used were: high, low, normal.
Time Frame: At Screening.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Screening time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 258
Percentage of participants
  RBC, Low | 3.9 | 2.7
  RBC, Normal | 84.4 | 81.8
  RBC, High | 11.7 | 15.5
  Neutrophils, Low | 12.8 | 10.9
  Neutrophils, Normal | 86.4 | 89.1
  Neutrophils, High | 0.8 | 0
  Lymphocytes, Low | 1.6 | 0
  Lymphocytes, Normal | 97.3 | 97.3
  Lymphocytes, High | 1.2 | 2.7
  WBC, Low | 3.5 | 1.2
  WBC, Normal | 94.9 | 97.3
  WBC, High | 1.6 | 1.6
  Haemoglobin, Low | 33.5 | 32.9
  Haemoglobin, Normal | 66.1 | 67.1
  Haemoglobin, High | 0.4 | 0
  Platelets, Low | 1.2 | 1.2
  Platelets, Normal | 80.2 | 77.5
  Platelets, High | 18.7 | 21.3

8. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: Haematological parameters assessed included: complete blood count (red blood cells [RBC], neutrophils, lymphocytes, white blood cells [WBC], haemoglobin, as well as differential count and platelet count for subjects aged 1-5 years, 6-12 years and 13-17 years. Reference range indicators used were: high, low, normal.
Time Frame: At Screening
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 89 | 91 | 68 | 67
Percentage of participants
  RBC, Low | 7.0 | 5.0 | 1.1 | 1.1 | 2.9 | 1.5
  RBC, Normal | 80.0 | 81.0 | 84.3 | 78.0 | 91.2 | 88.1
  RBC, High | 13.0 | 14.0 | 14.6 | 20.9 | 5.9 | 10.4
  Neutrophils, Low | 28.0 | 20.0 | 0 | 4.4 | 7.4 | 6.0
  Neutrophils, Normal | 72.0 | 80.0 | 97.8 | 95.6 | 92.6 | 94.0
  Neutrophils, High | 0 | 0 | 2.2 | 0 | 0 | 0
  Lymphocytes, Low | 0 | 0 | 0 | 0 | 5.9 | 0
  Lymphocytes, Normal | 98.0 | 95.0 | 100.0 | 97.8 | 92.6 | 100.0
  Lymphocytes, High | 2.0 | 5.0 | 0 | 2.2 | 1.5 | 0
  WBC, Low | 3.0 | 0 | 0 | 0 | 8.8 | 4.5
  WBC, Normal | 95.0 | 97.0 | 98.9 | 98.9 | 89.7 | 95.5
  WBC, High | 2.0 | 3.0 | 1.1 | 1.1 | 1.5 | 0
  Haemoglobin, Low | 38.0 | 36.0 | 14.6 | 14.3 | 51.5 | 53.7
  Haemoglobin, Normal | 62.0 | 64.0 | 85.4 | 85.7 | 47.1 | 46.3
  Haemoglobin, High | 0 | 0 | 0 | 0 | 1.5 | 0
  Platelets, Low | 0 | 0 | 0 | 0 | 4.4 | 4.5
  Platelets, Normal | 74.0 | 71.0 | 80.9 | 78.0 | 88.2 | 86.6
  Platelets, High | 26.0 | 29.0 | 19.1 | 22.0 | 7.4 | 9.0

9. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Day 3.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Day 3 time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 256
Percentage of participants
  RBC, Low | 5.1 | 6.3
  RBC, Normal | 86.8 | 82.4
  RBC, High | 8.2 | 11.3
  Neutrophils, Low | 28.4 | 11.7
  Neutrophils, Normal | 71.2 | 88.3
  Neutrophils, High | 0.4 | 0
  Lymphocytes, Low | 0.8 | 0
  Lymphocytes, Normal | 98.4 | 99.2
  Lymphocytes, High | 0.8 | 0.8
  WBC, Low | 7.8 | 2.3
  WBC, Normal | 90.7 | 96.1
  WBC, High | 1.6 | 1.6
  Haemoglobin, Low | 41.2 | 46.1
  Haemoglobin, Normal | 58.8 | 53.1
  Haemoglobin, High | 0 | 0.8
  Platelets, Low | 0.8 | 1.2
  Platelets, Normal | 87.5 | 82.4
  Platelets, High | 11.7 | 16.4

10. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Groups:
- GSK3390107A+Nimenrix 1-5YOAGroup: Sub-group of subjects from the GSK3390107A+Nimenrix Group, between and including 1 to 5 years of age (YOA), who received the investigational GSK3390107A vaccine at the Day 0 visit and Nimenrix at the Month 6 visit, intramuscularly into the thigh region.
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOAGroup | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 89 | 91 | 68 | 65
Percentage of participants
  RBC, Low | 6.0 | 9.0 | 2.2 | 4.4 | 7.4 | 4.6
  RBC, Normal | 82.0 | 80.0 | 89.9 | 82.4 | 89.7 | 86.2
  RBC, High | 12.0 | 11.0 | 7.9 | 13.2 | 2.9 | 9.2
  Neutrophils, Low | 47.0 | 22.0 | 14.6 | 4.4 | 19.1 | 6.2
  Neutrophils, Normal | 53.0 | 78.0 | 85.4 | 95.6 | 79.4 | 93.8
  Neutrophils, High | 0 | 0 | 0 | 0 | 1.5 | 0
  Lymphocytes, Low | 0 | 0 | 0 | 0 | 2.9 | 0
  Lymphocytes, Normal | 99.0 | 99.0 | 100.0 | 98.9 | 95.6 | 100.0
  Lymphocytes, High | 1.0 | 1.0 | 0 | 1.1 | 1.5 | 0
  WBC, Low | 6.0 | 2.0 | 4.5 | 2.2 | 14.7 | 3.1
  WBC, Normal | 92.0 | 94.0 | 95.5 | 97.8 | 82.4 | 96.9
  WBC, High | 2.0 | 4.0 | 0 | 0 | 2.9 | 0
  Haemoglobin, Low | 43.0 | 44.0 | 23.6 | 33.0 | 61.8 | 67.7
  Haemoglobin, Normal | 57.0 | 56.0 | 76.4 | 67.0 | 38.2 | 29.2
  Haemoglobin, High | 0 | 0 | 0 | 0 | 0 | 3.1
  Platelets, Low | 0 | 0 | 0 | 0 | 2.9 | 4.6
  Platelets, Normal | 79.0 | 77.0 | 93.3 | 84.6 | 92.6 | 87.7
  Platelets, High | 21.0 | 23.0 | 6.7 | 15.4 | 4.4 | 7.7

11. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Day 6.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Day 6 time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 256 | 256
Percentage of participants
  RBC, Low | 7.0 | 5.5
  RBC, Normal | 83.6 | 84.0
  RBC, High | 9.4 | 10.5
  Neutrophils, Low | 19.9 | 14.8
  Neutrophils, Normal | 79.3 | 84.8
  Neutrophils, High | 0.8 | 0.4
  Lymphocytes, Low | 1.2 | 0.8
  Lymphocytes, Normal | 97.7 | 97.3
  Lymphocytes, High | 1.2 | 2.0
  WBC, Low | 4.7 | 2.0
  WBC, Normal | 94.1 | 96.5
  WBC, High | 1.2 | 1.6
  Haemoglobin, Low | 42.6 | 44.1
  Haemoglobin, Normal | 57.4 | 55.1
  Haemoglobin, High | 0 | 0.8
  Platelets, Low | 2.3 | 2.0
  Platelets, Normal | 79.7 | 77.3
  Platelets, High | 18.0 | 20.7

12. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Day 6
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 99 | 98 | 89 | 91 | 68 | 67
Percentage of participants
  RBC, Low | 12.1 | 8.2 | 2.2 | 3.3 | 5.9 | 4.5
  RBC, Normal | 74.7 | 82.7 | 88.8 | 82.4 | 89.7 | 88.1
  RBC, High | 13.1 | 9.2 | 9.0 | 14.3 | 4.4 | 7.5
  Neutrophils, Low | 37.4 | 29.6 | 6.7 | 6.6 | 11.8 | 4.5
  Neutrophils, Normal | 61.6 | 69.4 | 92.1 | 93.4 | 88.2 | 95.5
  Neutrophils, High | 1.0 | 1.0 | 1.1 | 0 | 0 | 0
  Lymphocytes, Low | 1.0 | 0 | 0 | 0 | 2.9 | 3.0
  Lymphocytes, Normal | 97.0 | 95.9 | 98.9 | 98.9 | 97.1 | 97.0
  Lymphocytes, High | 2.0 | 4.1 | 1.1 | 1.1 | 0 | 0
  WBC, Low | 5.1 | 1.0 | 0 | 1.1 | 10.3 | 4.5
  WBC, Normal | 91.9 | 94.9 | 100.0 | 98.9 | 89.7 | 95.5
  WBC, High | 3.0 | 4.1 | 0 | 0 | 0 | 0
  Haemoglobin, Low | 50.5 | 40.8 | 22.5 | 36.3 | 57.4 | 59.7
  Haemoglobin, Normal | 49.5 | 59.2 | 77.5 | 63.7 | 42.6 | 37.3
  Haemoglobin, High | 0 | 0 | 0 | 0 | 0 | 3.0
  Platelets, Low | 0 | 0 | 0 | 0 | 8.8 | 7.5
  Platelets, Normal | 71.7 | 71.4 | 83.1 | 80.2 | 86.8 | 82.1
  Platelets, High | 28.3 | 28.6 | 16.9 | 19.8 | 4.4 | 10.4

13. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Day 30.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Day 30 time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 256
Percentage of participants
  RBC, Low | 4.7 | 3.5
  RBC, Normal | 83.7 | 82.4
  RBC, High | 11.7 | 14.1
  Neutrophils, Low | 18.3 | 15.6
  Neutrophils, Normal | 80.9 | 83.6
  Neutrophils, High | 0.8 | 0.8
  Lymphocytes, Low | 1.9 | 0.4
  Lymphocytes, Normal | 96.1 | 97.7
  Lymphocytes, High | 1.9 | 2.0
  WBC, Low | 5.4 | 3.1
  WBC, Normal | 93.0 | 95.3
  WBC, High | 1.6 | 1.6
  Haemoglobin, Low | 39.7 | 35.5
  Haemoglobin, Normal | 59.5 | 62.5
  Haemoglobin, High | 0.8 | 2.0
  Platelets, Low | 1.6 | 1.2
  Platelets, Normal | 87.9 | 84.0
  Platelets, High | 10.5 | 14.8

14. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Day 30
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 98 | 89 | 91 | 68 | 67
Percentage of participants
  RBC, Low | 9.0 | 6.1 | 2.2 | 2.2 | 1.5 | 1.5
  RBC, Normal | 73.0 | 75.5 | 88.8 | 85.7 | 92.6 | 88.1
  RBC, High | 18.0 | 18.4 | 9.0 | 12.1 | 5.9 | 10.4
  Neutrophils, Low | 35.0 | 30.6 | 11.2 | 5.5 | 2.9 | 7.5
  Neutrophils, Normal | 65.0 | 69.4 | 87.6 | 92.3 | 95.6 | 92.5
  Neutrophils, High | 0 | 0 | 1.1 | 2.2 | 1.5 | 0
  Lymphocytes, Low | 0 | 0 | 0 | 0 | 7.4 | 1.5
  Lymphocytes, Normal | 98.0 | 96.9 | 97.8 | 100.0 | 91.2 | 95.5
  Lymphocytes, High | 2.0 | 3.1 | 2.2 | 0 | 1.5 | 3.0
  WBC, Low | 5.0 | 3.1 | 4.5 | 3.3 | 7.4 | 3.0
  WBC, Normal | 94.0 | 95.9 | 93.3 | 95.6 | 91.2 | 94.0
  WBC, High | 1.0 | 1.0 | 2.2 | 1.1 | 1.5 | 3.0
  Haemoglobin, Low | 37.0 | 31.6 | 38.2 | 35.2 | 45.6 | 41.8
  Haemoglobin, Normal | 62.0 | 67.3 | 61.8 | 64.8 | 52.9 | 52.2
  Haemoglobin, High | 1.0 | 1.0 | 0 | 0 | 1.5 | 6.0
  Platelets, Low | 0 | 0 | 0 | 0 | 5.9 | 4.5
  Platelets, Normal | 82.0 | 82.7 | 93.3 | 85.7 | 89.7 | 83.6
  Platelets, High | 18.0 | 17.3 | 6.7 | 14.3 | 4.4 | 11.9

15. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Month 6.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Month 6 time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 254
Percentage of participants
  RBC, Low | 7.8 | 6.7
  RBC, Normal | 80.5 | 81.5
  RBC, High | 11.7 | 11.8
  Neutrophils, Low | 21.0 | 17.7
  Neutrophils, Normal | 79.0 | 81.1
  Neutrophils, High | 0 | 1.2
  Lymphocytes, Low | 0.4 | 0
  Lymphocytes, Normal | 97.7 | 97.6
  Lymphocytes, High | 1.9 | 2.4
  WBC, Low | 7.4 | 3.5
  WBC, Normal | 92.2 | 93.7
  WBC, High | 0.4 | 2.8
  Haemoglobin, Low | 38.1 | 34.3
  Haemoglobin, Normal | 61.9 | 65.7
  Haemoglobin, High | 0 | 0
  Platelets, Low | 0.8 | 0
  Platelets, Normal | 88.7 | 85.8
  Platelets, High | 10.5 | 14.2

16. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Month 6
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 96 | 89 | 91 | 68 | 67
Percentage of participants
  RBC, Low | 16.0 | 15.6 | 2.2 | 1.1 | 2.9 | 1.5
  RBC, Normal | 78.0 | 76.0 | 78.7 | 78.0 | 86.8 | 94.0
  RBC, High | 6.0 | 8.3 | 19.1 | 20.9 | 10.3 | 4.5
  Neutrophils, Low | 38.0 | 28.1 | 7.9 | 12.1 | 13.2 | 10.4
  Neutrophils, Normal | 62.0 | 70.8 | 92.1 | 85.7 | 86.8 | 89.6
  Neutrophils, High | 0 | 1.0 | 0 | 2.2 | 0 | 0
  Lymphocytes, Low | 0 | 0 | 0 | 0 | 1.5 | 0
  Lymphocytes, Normal | 96.0 | 96.9 | 100.0 | 97.8 | 97.1 | 98.5
  Lymphocytes, High | 4.0 | 3.1 | 0 | 2.2 | 1.5 | 1.5
  WBC, Low | 6.0 | 4.2 | 3.4 | 2.2 | 14.7 | 4.5
  WBC, Normal | 93.0 | 92.7 | 96.6 | 94.5 | 85.3 | 94.0
  WBC, High | 1.0 | 3.1 | 0 | 3.3 | 0 | 1.5
  Haemoglobin, Low | 51.0 | 43.8 | 21.3 | 22.0 | 41.2 | 37.3
  Haemoglobin, Normal | 49.0 | 56.3 | 78.7 | 78.0 | 58.8 | 62.7
  Haemoglobin, High | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, Low | 0 | 0 | 0 | 0 | 2.9 | 0
  Platelets, Normal | 89.0 | 87.5 | 87.6 | 85.7 | 89.7 | 83.6
  Platelets, High | 11.0 | 12.5 | 12.4 | 14.3 | 7.4 | 16.4

17. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Month 6 + 6 Days.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Month 6 + 6 Days time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 253 | 250
Percentage of participants
  RBC, Low | 7.5 | 5.6
  RBC, Normal | 84.6 | 83.6
  RBC, High | 7.9 | 10.8
  Neutrophils, Low | 20.9 | 28.8
  Neutrophils, Normal | 78.7 | 71.2
  Neutrophils, High | 0.4 | 0
  Lymphocytes, Low | 0 | 0
  Lymphocytes, Normal | 99.2 | 98.0
  Lymphocytes, High | 0.8 | 2.0
  WBC, Low | 4.3 | 7.6
  WBC, Normal | 94.5 | 90.8
  WBC, High | 1.2 | 1.6
  Haemoglobin, Low | 38.7 | 41.6
  Haemoglobin, Normal | 60.9 | 58.4
  Haemoglobin, High | 0.4 | 0
  Platelets, Low | 0.4 | 1.2
  Platelets, Normal | 87.4 | 81.6
  Platelets, High | 12.3 | 17.2

18. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Month 6 + 6 Days
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 98 | 93 | 89 | 90 | 66 | 67
Percentage of participants
  RBC, Low | 18.4 | 14.0 | 0 | 1.1 | 1.5 | 0
  RBC, Normal | 77.6 | 78.5 | 87.6 | 81.1 | 90.9 | 94.0
  RBC, High | 4.1 | 7.5 | 12.4 | 17.8 | 7.6 | 6.0
  Neutrophils, Low | 44.9 | 48.4 | 5.6 | 18.9 | 6.1 | 14.9
  Neutrophils, Normal | 55.1 | 51.6 | 93.3 | 81.1 | 93.9 | 85.1
  Neutrophils, High | 0 | 0 | 1.1 | 0 | 0 | 0
  Lymphocytes, Low | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Normal | 98.0 | 96.8 | 100.0 | 97.8 | 100.0 | 100.0
  Lymphocytes, High | 2.0 | 3.2 | 0 | 2.2 | 0 | 0
  WBC, Low | 5.1 | 6.5 | 1.1 | 6.7 | 7.6 | 10.4
  WBC, Normal | 91.8 | 91.4 | 98.9 | 91.1 | 92.4 | 89.6
  WBC, High | 3.1 | 2.2 | 0 | 2.2 | 0 | 0
  Haemoglobin, Low | 56.1 | 51.6 | 19.1 | 27.8 | 39.4 | 46.3
  Haemoglobin, Normal | 43.9 | 48.4 | 80.9 | 72.2 | 59.1 | 53.7
  Haemoglobin, High | 0 | 0 | 0 | 0 | 1.5 | 0
  Platelets, Low | 0 | 0 | 0 | 0 | 1.5 | 4.5
  Platelets, Normal | 88.8 | 81.7 | 85.4 | 80.0 | 87.9 | 83.6
  Platelets, High | 11.2 | 18.3 | 14.6 | 20.0 | 10.6 | 11.9

19. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Month 6 + 30 Days.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Month 6 + 30 Days time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 254 | 250
Percentage of participants
  RBC, Low | 4.7 | 4.4
  RBC, Normal | 81.9 | 83.6
  RBC, High | 13.4 | 12.0
  Neutrophils, Low | 24.4 | 25.6
  Neutrophils, Normal | 75.6 | 73.2
  Neutrophils, High | 0 | 1.2
  Lymphocytes, Low | 0.8 | 0.8
  Lymphocytes, Normal | 98.0 | 98.0
  Lymphocytes, High | 1.2 | 1.2
  WBC, Low | 5.5 | 6.4
  WBC, Normal | 93.7 | 92.8
  WBC, High | 0.8 | 0.8
  Haemoglobin, Low | 35.0 | 37.6
  Haemoglobin, Normal | 65.0 | 62.0
  Haemoglobin, High | 0 | 0.4
  Platelets, Low | 0.4 | 1.6
  Platelets, Normal | 86.2 | 85.2
  Platelets, High | 13.4 | 13.2

20. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Month 6 + 30 Days
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 98 | 93 | 89 | 90 | 67 | 67
Percentage of participants
  RBC, Low | 9.2 | 11.8 | 2.2 | 0 | 1.5 | 0
  RBC, Normal | 76.5 | 74.2 | 82.0 | 86.7 | 89.6 | 92.5
  RBC, High | 14.3 | 14.0 | 15.7 | 13.3 | 9.0 | 7.5
  Neutrophils, Low | 52.0 | 57.0 | 10.1 | 8.9 | 3.0 | 4.5
  Neutrophils, Normal | 48.0 | 43.0 | 89.9 | 87.8 | 97.0 | 95.5
  Neutrophils, High | 0 | 0 | 0 | 3.3 | 0 | 0
  Lymphocytes, Low | 0 | 0 | 1.1 | 1.1 | 1.5 | 1.5
  Lymphocytes, Normal | 98.0 | 97.8 | 98.9 | 98.9 | 97.0 | 97.0
  Lymphocytes, High | 2.0 | 2.2 | 0 | 0 | 1.5 | 1.5
  WBC, Low | 7.1 | 7.5 | 3.4 | 6.7 | 6.0 | 4.5
  WBC, Normal | 90.8 | 92.5 | 96.6 | 92.2 | 94.0 | 94.0
  WBC, High | 2.0 | 0 | 0 | 1.1 | 0 | 1.5
  Haemoglobin, Low | 44.9 | 37.6 | 24.7 | 28.9 | 34.3 | 49.3
  Haemoglobin, Normal | 55.1 | 62.4 | 75.3 | 71.1 | 65.7 | 49.3
  Haemoglobin, High | 0 | 0 | 0 | 0 | 0 | 1.5
  Platelets, Low | 0 | 2.2 | 1.1 | 2.2 | 0 | 0
  Platelets, Normal | 84.7 | 86.0 | 86.5 | 87.8 | 88.1 | 80.6
  Platelets, High | 15.3 | 11.8 | 12.4 | 10.0 | 11.9 | 19.4

21. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, Overall
Description: as for outcome 7
Time Frame: At Month 12.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with available results at the Month 12 time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 253 | 254
Percentage of participants
  RBC, Low | 6.3 | 10.2
  RBC, Normal | 83.0 | 81.1
  RBC, High | 10.7 | 8.7
  Neutrophils, Low | 22.1 | 18.5
  Neutrophils, Normal | 77.9 | 81.5
  Neutrophils, High | 0 | 0
  Lymphocytes, Low | 0.4 | 0.8
  Lymphocytes, Normal | 99.2 | 97.6
  Lymphocytes, High | 0.4 | 1.6
  WBC, Low | 6.3 | 4.7
  WBC, Normal | 92.9 | 93.3
  WBC, High | 0.8 | 2.0
  Haemoglobin, Low | 42.7 | 46.1
  Haemoglobin, Normal | 56.9 | 53.9
  Haemoglobin, High | 0.4 | 0
  Platelets, Low | 0.8 | 1.2
  Platelets, Normal | 87.0 | 83.9
  Platelets, High | 12.3 | 15.0

22. Primary Outcome: Percentage of Subjects With Haematological Laboratory Abnormalities, by Age Stratum
Description: as for outcome 8
Time Frame: At Month 12
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 97 | 88 | 90 | 65 | 67
Percentage of participants
  RBC, Low | 13.0 | 23.7 | 3.4 | 0 | 0 | 4.5
  RBC, Normal | 74.0 | 64.9 | 86.4 | 88.9 | 92.3 | 94.0
  RBC, High | 13.0 | 11.3 | 10.2 | 11.1 | 7.7 | 1.5
  Neutrophils, Low | 47.0 | 40.2 | 2.3 | 6.7 | 10.8 | 3.0
  Neutrophils, Normal | 53.0 | 59.8 | 97.7 | 93.3 | 89.2 | 97.0
  Neutrophils, High | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, Low | 1.0 | 0 | 0 | 1.1 | 0 | 1.5
  Lymphocytes, Normal | 98.0 | 96.9 | 100.0 | 97.8 | 100.0 | 98.5
  Lymphocytes, High | 1.0 | 3.1 | 0 | 1.1 | 0 | 0
  WBC, Low | 5.0 | 8.2 | 3.4 | 2.2 | 12.3 | 3.0
  WBC, Normal | 93.0 | 86.6 | 96.6 | 97.8 | 87.7 | 97.0
  WBC, High | 2.0 | 5.2 | 0 | 0 | 0 | 0
  Haemoglobin, Low | 50.0 | 53.6 | 31.8 | 32.2 | 46.2 | 53.7
  Haemoglobin, Normal | 50.0 | 46.4 | 68.2 | 67.8 | 52.3 | 46.3
  Haemoglobin, High | 0 | 0 | 0 | 0 | 1.5 | 0
  Platelets, Low | 1.0 | 2.1 | 0 | 0 | 1.5 | 1.5
  Platelets, Normal | 82.0 | 80.4 | 86.4 | 85.6 | 95.4 | 86.6
  Platelets, High | 17.0 | 17.5 | 13.6 | 14.4 | 3.1 | 11.9

23. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: Biochemical parameters assessed included: alanine aminotransferase [ALT], creatinine [CRE] for all subjects, in both groups. Reference range indicators used were: high, low, normal.
Time Frame: At Screening.
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 258
Percentage of participants
  ALT, Low | 24.1 | 29.1
  ALT, Normal | 75.1 | 70.5
  ALT, High | 0.8 | 0.4
  CRE, Low | 3.5 | 2.3
  CRE, Normal | 89.9 | 92.2
  CRE, High | 6.6 | 5.4

24. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: Biochemical parameters assessed included: alanine aminotransferase [ALT], creatinine [CRE] for subjects aged 1-5 years, 6-12 years and 13-17 years. Reference range indicators used were: high, low, normal.
Time Frame: At Screening
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 89 | 91 | 68 | 67
Percentage of participants
  ALT, Low | 24.0 | 35.0 | 27.0 | 27.5 | 20.6 | 22.4
  ALT, Normal | 76.0 | 65.0 | 70.8 | 71.4 | 79.4 | 77.6
  ALT, High | 0 | 0 | 2.2 | 1.1 | 0 | 0
  CRE, Low | 2.0 | 3.0 | 0 | 0 | 10.3 | 4.5
  CRE, Normal | 83.0 | 84.0 | 97.8 | 98.9 | 89.7 | 95.5
  CRE, High | 15.0 | 13.0 | 2.2 | 1.1 | 0 | 0

25. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Day 3.
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 257
Percentage of participants
  ALT, Low | 26.1 | 29.6
  ALT, Normal | 73.5 | 69.3
  ALT, High | 0.4 | 1.2
  CRE, Low | 1.2 | 1.6
  CRE, Normal | 93.4 | 90.7
  CRE, High | 5.4 | 7.8

26. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Day 3
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 89 | 91 | 68 | 66
Percentage of participants
  ALT, Low | 31.0 | 43.0 | 28.1 | 23.1 | 16.2 | 18.2
  ALT, Normal | 69.0 | 57.0 | 71.9 | 74.7 | 82.4 | 80.3
  ALT, High | 0 | 0 | 0 | 2.2 | 1.5 | 1.5
  CRE, Low | 1.0 | 3.0 | 0 | 0 | 2.9 | 1.5
  CRE, Normal | 85.0 | 78.0 | 100.0 | 98.9 | 97.1 | 98.5
  CRE, High | 14.0 | 19.0 | 0 | 1.1 | 0 | 0

27. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Day 6.
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 256 | 256
Percentage of participants
  ALT, Low | 27.7 | 29.3
  ALT, Normal | 71.9 | 69.9
  ALT, High | 0.4 | 0.8
  CRE, Low | 2.7 | 2.0
  CRE, Normal | 89.5 | 93.4
  CRE, High | 7.8 | 4.7

28. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Day 6
Population: as for outcome 11
Measure: Number; unit: Percentage of particcipants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 99 | 98 | 89 | 91 | 68 | 67
Percentage of particcipants
  ALT, Low | 31.3 | 39.8 | 25.8 | 24.2 | 25.0 | 20.9
  ALT, Normal | 68.7 | 60.2 | 74.2 | 74.7 | 73.5 | 77.6
  ALT, High | 0 | 0 | 0 | 1.1 | 1.5 | 1.5
  CRE, Low | 2.0 | 2.0 | 0 | 0 | 7.4 | 4.5
  CRE, Normal | 77.8 | 85.7 | 100.0 | 100.0 | 92.6 | 95.5
  CRE, High | 20.2 | 12.2 | 0 | 0 | 0 | 0

29. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Day 30.
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 256
Percentage of participants
  ALT, Low | 29.6 | 28.9
  ALT, Normal | 70.0 | 71.1
  ALT, High | 0.4 | 0
  CRE, Low | 2.3 | 2.0
  CRE, Normal | 90.3 | 89.5
  CRE, High | 7.4 | 8.6

30. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Day 30
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 98 | 89 | 91 | 68 | 67
Percentage of participants
  ALT, Low | 30.0 | 40.8 | 33.7 | 29.7 | 23.5 | 10.4
  ALT, Normal | 70.0 | 59.2 | 65.2 | 70.3 | 76.5 | 89.6
  ALT, High | 0 | 0 | 1.1 | 0 | 0 | 0
  CRE, Low | 1.0 | 3.1 | 0 | 1.1 | 7.4 | 1.5
  CRE, Normal | 82.0 | 75.5 | 100.0 | 98.9 | 89.7 | 97.0
  CRE, High | 17.0 | 21.4 | 0 | 0 | 2.9 | 1.5

31. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Month 6.
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 257 | 254
Percentage of participants
  ALT, Low | 20.2 | 15.4
  ALT, Normal | 79.4 | 84.3
  ALT, High | 0.4 | 0.4
  CRE, Low | 14.0 | 13.0
  CRE, Normal | 84.4 | 86.6
  CRE, High | 1.6 | 0.4

32. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Month 6
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 96 | 89 | 91 | 68 | 67
Percentage of participants
  ALT, Low | 18.0 | 20.8 | 12.4 | 8.8 | 33.8 | 16.4
  ALT, Normal | 82.0 | 78.1 | 86.5 | 91.2 | 66.2 | 83.6
  ALT, High | 0 | 1.0 | 1.1 | 0 | 0 | 0
  CRE, Low | 27.0 | 22.9 | 0 | 0 | 13.2 | 16.4
  CRE, Normal | 70.0 | 76.0 | 100.0 | 100.0 | 85.3 | 83.6
  CRE, High | 3.0 | 1.0 | 0 | 0 | 1.5 | 0

33. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Month 6 + 6 Days.
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 253 | 250
Percentage of participants
  ALT, Low | 19.8 | 22.4
  ALT, Normal | 79.1 | 77.6
  ALT, High | 1.2 | 0
  CRE, Low | 13.8 | 13.2
  CRE, Normal | 85.4 | 86.4
  CRE, High | 0.8 | 0.4

34. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Month 6 + 6 Days
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 98 | 93 | 89 | 90 | 66 | 67
Percentage of participants
  ALT, Low | 17.3 | 28.0 | 14.6 | 17.8 | 30.3 | 20.9
  ALT, Normal | 81.6 | 72.0 | 83.1 | 82.2 | 69.7 | 79.1
  ALT, High | 1.0 | 0 | 2.2 | 0 | 0 | 0
  CRE, Low | 26.5 | 29.0 | 2.2 | 0 | 10.6 | 9.0
  CRE, Normal | 71.4 | 71.0 | 97.8 | 98.9 | 89.4 | 91.0
  CRE, High | 2.0 | 0 | 0 | 1.1 | 0 | 0

35. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Month 6 + 30 Days.
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 254 | 250
Percentage of participants
  ALT, Low | 15.7 | 17.2
  ALT, Normal | 82.3 | 81.2
  ALT, High | 2.0 | 1.6
  CRE, Low | 15.4 | 15.2
  CRE, Normal | 83.1 | 83.6
  CRE, High | 1.6 | 1.2

36. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Month 6 + 30 Days
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 98 | 93 | 89 | 90 | 67 | 67
Percentage of participants
  ALT, Low | 14.3 | 17.2 | 10.1 | 13.3 | 25.4 | 22.4
  ALT, Normal | 82.7 | 82.8 | 87.6 | 83.3 | 74.6 | 76.1
  ALT, High | 3.1 | 0 | 2.2 | 3.3 | 0 | 1.5
  CRE, Low | 27.6 | 33.3 | 2.2 | 0 | 14.9 | 10.4
  CRE, Normal | 71.4 | 66.7 | 95.5 | 96.7 | 83.6 | 89.6
  CRE, High | 1.0 | 0 | 2.2 | 3.3 | 1.5 | 0

37. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, Overall
Description: as for outcome 23
Time Frame: At Month 12.
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 253 | 254
Percentage of participants
  ALT, Low | 32.4 | 26.4
  ALT, Normal | 66.8 | 72.0
  ALT, High | 0.8 | 1.6
  CRE, Low | 15.4 | 15.0
  CRE, Normal | 77.1 | 79.5
  CRE, High | 7.5 | 5.5

38. Primary Outcome: Percentage of Subjects With Biochemical Laboratory Abnormalities, by Age Stratum
Description: as for outcome 24
Time Frame: At Month 12
Population: as for outcome 21
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 97 | 88 | 90 | 65 | 67
Percentage of participants
  ALT, Low | 26.0 | 27.8 | 39.8 | 25.6 | 32.3 | 25.4
  ALT, Normal | 73.0 | 71.1 | 59.1 | 74.4 | 67.7 | 70.1
  ALT, High | 1.0 | 1.0 | 1.1 | 0 | 0 | 4.5
  CRE, Low | 21.0 | 18.6 | 6.8 | 7.8 | 18.5 | 19.4
  CRE, Normal | 73.0 | 77.3 | 79.5 | 83.3 | 80.0 | 77.6
  CRE, High | 6.0 | 4.1 | 13.6 | 8.9 | 1.5 | 3.0

39. Primary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESI), Overall
Description: AESI included clinical symptoms of thrombocytopenia for all subjects, in both groups.
Time Frame: During the 7 day follow-up period after vaccination at Day 0 (i.e., Day 0 up to Day 6)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 300 | 300
Participants | 0 | 0

40. Primary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESI), by Age Stratum
Description: AESI included clinical symptoms of thrombocytopenia for subjects aged 1-5 years, 6-12 years and 13-17 years.
Time Frame: During the 7 day follow-up period after vaccination at Day 0 (i.e. Day 0 up to Day 6)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 99 | 101 | 101 | 99
Participants | 0 | 0 | 0 | 0 | 0 | 0

41. Primary Outcome: Number of Subjects With Serious Adverse Events, Overall
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. SAEs, for this endpoint, were assessed in all subjects, in both groups.
Time Frame: During the entire study period: From Screening to Month 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 300 | 300
Participants | 2 | 2

42. Primary Outcome: Number of Subjects With Serious Adverse Events, by Age Stratum
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. SAEs, for this endpoint, were assessed in subjects aged 1-5 years, 6-12 years and 13-17 years.
Time Frame: During the entire study period: From Screening to Month 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 99 | 101 | 101 | 99
Participants | 0 | 1 | 1 | 1 | 1 | 0

43. Secondary Outcome: Anti-glycoprotein (GP) Ebola Virus Zaire (EBOV) Antibody Titers, Overall
Description: Anti-GP EBOV antibodies were expressed as Geometric Mean Titers (GMTs), as measured by the Enzyme-Linked Immunosorbent Assay (ELISA) and assessed in all subjects, in both groups.
Time Frame: At Day 0, Day 30, Month 6, Month 6 + 30 Days and Month 12.
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for analysis of immunogenicity, which included all evaluable subjects who complied with the protocol requirements and procedures and for whom data concerning immunogenicity endpoint measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 295 | 294
Titers
  Anti-GP EBOV, Day 0 | 24.755 [22.673 to 27.029] | 24.587 [22.612 to 26.735]
  Anti-GP EBOV, Day 30: number analyzed (Participants) | 243 | 238
  Anti-GP EBOV, Day 30 | 1739.756 [1562.966 to 1936.543] | 24.372 [22.236 to 26.714]
  Anti-GP EBOV, Month 6: number analyzed (Participants) | 240 | 234
  Anti-GP EBOV, Month 6 | 1017.712 [925.011 to 1119.702] | 23.343 [21.616 to 25.208]
  Anti-GP EBOV, Month 6 + Day 30: number analyzed (Participants) | 240 | 234
  Anti-GP EBOV, Month 6 + Day 30 | 970.870 [883.886 to 1066.414] | 1513.928 [1370.915 to 1671.859]
  Anti-GP EBOV, Month 12: number analyzed (Participants) | 238 | 235
  Anti-GP EBOV, Month 12 | 909.092 [813.891 to 1015.429] | 889.641 [800.009 to 989.315]

44. Secondary Outcome: Anti-GP EBOV Antibody Titers, by Age Stratum
Description: Anti-GP EBOV antibodies were expressed as Geometric Mean Titers (GMTs), as measured by the Enzyme-Linked Immunosorbent Assay (ELISA) and assessed in subjects aged 1-5 years, 6-12 years and 13-17 years.
Time Frame: At Day 0, Day 30, Month 6, Month 6 + 30 Days and Month 12
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 96 | 98 | 99 | 96
Titers
  Anti-GP EBOV, Day 0 | 29.526 [24.175 to 36.062] | 31.545 [26.543 to 37.489] | 22.764 [20.195 to 25.661] | 21.241 [18.973 to 23.780] | 22.473 [19.966 to 25.295] | 22.021 [19.281 to 25.151]
  Anti-GP EBOV, Day 30: number analyzed (Participants) | 77 | 65 | 82 | 89 | 84 | 84
  Anti-GP EBOV, Day 30 | 1564.283 [1339.748 to 1826.449] | 29.565 [24.794 to 35.254] | 1394.540 [1174.847 to 1655.316] | 21.879 [19.098 to 25.065] | 2405.635 [1942.446 to 2979.274] | 22.300 [18.991 to 26.186]
  Anti-GP EBOV, Month 6: number analyzed (Participants) | 77 | 64 | 82 | 89 | 81 | 81
  Anti-GP EBOV, Month 6 | 705.913 [619.567 to 804.292] | 23.328 [20.814 to 26.146] | 1030.880 [887.724 to 1197.121] | 21.834 [19.476 to 24.478] | 1482.304 [1231.572 to 1784.081] | 25.141 [21.161 to 29.871]
  Anti-GP EBOV, Month 6 + 30 Days: number analyzed (Participants) | 76 | 63 | 82 | 89 | 82 | 82
  Anti-GP EBOV, Month 6 + 30 Days | 722.550 [638.466 to 817.708] | 1150.199 [971.093 to 1362.339] | 885.295 [766.161 to 1022.954] | 1399.458 [1188.609 to 1647.710] | 1439.460 [1193.726 to 1735.780] | 2190.763 [1862.359 to 2577.076]
  Anti-GP EBOV, Month 12: number analyzed (Participants) | 77 | 64 | 81 | 89 | 80 | 82
  Anti-GP EBOV, Month 12 | 715.890 [619.208 to 827.668] | 583.371 [486.760 to 699.158] | 751.765 [645.194 to 875.939] | 883.668 [759.207 to 1028.533] | 1424.270 [1118.513 to 1813.608] | 1412.293 [1179.201 to 1691.459]

45. Secondary Outcome: Percentage of Seronegative/Seropositive Subjects for Anti-GP EBOV Antibodies, Overall
Description: A seronegative subject is a subject whose titer is below the cut-off value. A seropositive subject is a subject whose titer is greater than or equal to the cut-off value. The analysis, for this endpoint, was performed on all subjects, in both groups.
Time Frame: At Day 0, Day 30, Month 6 and Month 6 + 30 Days.
Population: as for outcome 43
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
Number analyzed (Participants) | 295 | 294
Percentage of participants
  Anti-GP EBOV, Day 0, S- | 82.7 | 82.3
  Anti-GP EBOV, Day 0, S+ | 17.3 | 17.7
  Anti-GP EBOV, Day 30, S-: number analyzed (Participants) | 293 | 290
  Anti-GP EBOV, Day 30, S- | 0.7 | 83.8
  Anti-GP EBOV, Day 30, S+: number analyzed (Participants) | 293 | 290
  Anti-GP EBOV, Day 30, S+ | 99.3 | 16.2
  Anti-GP EBOV, Month 6, S-: number analyzed (Participants) | 290 | 282
  Anti-GP EBOV, Month 6, S- | 0.0 | 84.0
  Anti-GP EBOV, Month 6, S+: number analyzed (Participants) | 290 | 282
  Anti-GP EBOV, Month 6, S+ | 100.0 | 16.0
  Anti-GP EBOV, Month 6 + 30 Days, S-: number analyzed (Participants) | 290 | 281
  Anti-GP EBOV, Month 6 + 30 Days, S- | 0.0 | 0.0
  Anti-GP EBOV, Month 6 + 30 Days, S+: number analyzed (Participants) | 290 | 281
  Anti-GP EBOV, Month 6 + 30 Days, S+ | 100.0 | 100.0

46. Secondary Outcome: Percentage of Seronegative/Seropositive Subjects for Anti-GP EBOV Antibodies, by Age Stratum
Description: A seronegative subject is a subject whose titer is below the cut-off value. A seropositive subject is a subject whose titer is greater than or equal to the cut-off value. The analysis, for this endpoint, was performed on subjects aged 1-5 years, 6-12 years and 13-17 years.
Time Frame: At Day 0, Day 30, Month 6 and Month 6 + 30 Days
Population: as for outcome 43
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3390107A+Nimenrix 13-17YOA Group | Nimenrix+GSK3390107A 13-17YOA Group | GSK3390107A+Nimenrix 6-12YOA Group | Nimenrix+GSK3390107A 6-12YOA Group | GSK3390107A+Nimenrix 1-5YOA Group | Nimenrix+GSK3390107A 1-5YOA Group
Number analyzed (Participants) | 100 | 100 | 96 | 98 | 99 | 96
Percentage of participants
  Anti-GP EBOV, Day 0, S- | 77.0 | 67.0 | 85.4 | 90.8 | 85.9 | 89.6
  Anti-GP EBOV, Day 0, S+ | 23.0 | 33.0 | 14.6 | 9.2 | 14.1 | 10.4
  Anti-GP EBOV, Day 30, S-: number analyzed (Participants) | 99 | 98 | 96 | 98 | 98 | 94
  Anti-GP EBOV, Day 30, S- | 0 | 70.4 | 0 | 90.8 | 2.0 | 90.4
  Anti-GP EBOV, Day 30, S+: number analyzed (Participants) | 99 | 98 | 96 | 98 | 98 | 94
  Anti-GP EBOV, Day 30, S+ | 100.0 | 29.6 | 100.0 | 9.2 | 98.0 | 9.6
  Anti-GP EBOV, Month 6, S-: number analyzed (Participants) | 100 | 95 | 96 | 98 | 94 | 89
  Anti-GP EBOV, Month 6, S- | 0 | 80.0 | 0 | 88.8 | 0 | 83.1
  Anti-GP EBOV, Month 6, S+: number analyzed (Participants) | 100 | 95 | 96 | 98 | 94 | 89
  Anti-GP EBOV, Month 6, S+ | 100.0 | 20.0 | 100.0 | 11.2 | 100.0 | 16.9
  Anti-GP EBOV, Month 6 + 30 Days, S-: number analyzed (Participants) | 98 | 93 | 96 | 98 | 96 | 90
  Anti-GP EBOV, Month 6 + 30 Days, S- | 0 | 0 | 0 | 0 | 0 | 0
  Anti-GP EBOV, Month 6 + 30 Days, S+: number analyzed (Participants) | 98 | 93 | 96 | 98 | 96 | 90
  Anti-GP EBOV, Month 6 + 30 Days, S+ | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: from Screening up to study end at Month 12.
Description: From Screening to Day 0, only those SAEs that were considered related to study participation or to concurrent use of GlaxoSmithKline (GSK) medication/ vaccine needed to be recorded.
Arm/Group | GSK3390107A+Nimenrix Group | Nimenrix+GSK3390107A Group
All-Cause Mortality (participants affected / at risk) | 1/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 2/300 | 3/300
Other Adverse Events (participants affected / at risk) | 194/300 | 89/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3390107A+Nimenrix Group (N=300) | Nimenrix+GSK3390107A Group (N=300)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS D (Infections and infestations) | 0 (0) | 1 (1)
MALARIA (Infections and infestations) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3390107A+Nimenrix Group (N=300) | Nimenrix+GSK3390107A Group (N=300)
PAIN (General disorders) | 127 (189) | 60 (82)
PYREXIA (General disorders) | 95 (112) | 28 (37)
FATIGUE (General disorders) | 33 (37) | 6 (8)
HEADACHE (Nervous system disorders) | 62 (72) | 17 (19)
SOMNOLENCE (Nervous system disorders) | 26 (37) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 (32) | 4 (6)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 16 (22) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02548078/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02548078/SAP_001.pdf